CLINICAL TRIAL: NCT06995846
Title: Application of Bacterial DNA Quantitative Detection in Diagnosis of SBP in Cirrhosis: A Multi Center Diagnostic Experiment
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Zhongjie Hu, associate dean, Beijing YouAn Hospital
Other Study IDs: LL-2024-034-K
Record Dates: First submitted 2025-05-28; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis; Ascites; Bacterial Infections
MeSH Terms: conditions — Fibrosis; Ascites; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic Patients with Ascites: Cirrhotic Patients with Ascites
  Interventions: Diagnostic Test: Bacterial DNA Levels in Ascites

INTERVENTIONS:
Diagnostic Test: Bacterial DNA Levels in Ascites — The bactDNA was detected by droplet digital polymerase chain reaction (ddPCR).

SUMMARY:
Background and Significance:

Spontaneous bacterial peritonitis (SBP) is a common and life-threatening complication in patients with liver cirrhosis, characterized by high incidence and mortality. The current diagnostic standard relies on ascitic fluid polymorphonuclear leukocyte (PMN) count ≥250 cells/μL. However, this threshold is associated with high rates of missed diagnoses, poor correlation with clinical symptoms, and delays in pathogen identification due to the low sensitivity and prolonged time of traditional ascitic fluid culture.

With the development of molecular diagnostics, bacterial DNA (bactDNA) detection-especially through droplet digital PCR (ddPCR)-has emerged as a promising technique due to its high sensitivity, absolute quantification capability, and robustness. This study aims to evaluate the diagnostic value and accuracy of ddPCR-based quantification of bacterial DNA in ascitic fluid for SBP, providing a novel and objective diagnostic tool to improve early and accurate detection and to inform targeted antimicrobial therapy.

Objectives:

To assess the diagnostic accuracy (sensitivity, specificity, predictive values) of ddPCR-based quantification of total bacterial DNA in ascitic fluid for SBP.

To evaluate the diagnostic performance of the ratio of Gram-positive to Gram-negative bacterial DNA (G+/G-) in predicting SBP.

To explore the potential of ddPCR-based bacterial DNA quantification as a complementary or alternative method to conventional PMN-based diagnostic criteria.

Study Design and Methods:

This is a prospective diagnostic study involving 700 patients with liver cirrhosis and ascites. Ascitic fluid samples will be analyzed using ddPCR to quantify bacterial DNA levels. These results will be compared with traditional diagnostic criteria, including PMN counts and expert panel assessments based on clinical symptoms and laboratory findings. Statistical analyses will include correlation analysis, ROC curve analysis, and consistency testing.

Expected Outcomes:

The study aims to establish the clinical efficacy of ddPCR-based quantification of bacterial DNA in ascitic fluid as a novel diagnostic marker for SBP. This method is expected to be particularly useful in atypical cases where PMN counts are <250/μL and may help guide preliminary antibiotic selection based on the proportion of Gram-positive and Gram-negative bacteria, thereby reducing empirical treatment failures and antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no restriction on gender.
* Diagnosis of liver cirrhosis based on imaging, biochemical, or hematological evidence of impaired hepatic synthetic function or portal hypertension, or histologically confirmed cirrhosis, regardless of etiology.
* Diagnosis of ascites according to the 2023 Chinese Clinical Guidelines for the Diagnosis and Treatment of Cirrhotic Ascites and Related Complications.

Exclusion Criteria:

* Patients with confirmed infections in other tissues or organs.
* Ascites caused by non-hepatic etiologies, such as renal or cardiac ascites.
* Pregnant individuals, intravenous drug users, or HIV-infected individuals.
* Patients with uncontrolled hepatocellular carcinoma or other systemic malignancies.
* Patients who have previously undergone organ transplantation.
* Patients currently receiving glucocorticoids or other immunosuppressive therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic ascites patients admitted to the liver disease departments of our hospital and various sub centers
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
spontaneous bacterial peritonitis (SBP) | From enrollment to the end of follow at 24 weeks
  The SBP diagnosis is based on PMN (2021 practice Guidelines on the management of ascites in cirrhosis.) a clinical composite diagnosis (2023 Chinese guidelines)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 8 You An Men Wai Street, Fengtai District, Beijing 100069, China, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial